CLINICAL TRIAL: NCT01834495
Title: Phase 4 Study of Efficacy of Balloon-Expandable Cobalt Chromium SCUBA Stent Versus Self-Expandable Stent COMPLETE-SE Nitinol Stenting for the Atherosclerotic ILIAC Arterial Disease: Prospective, Multicenter, Randomized, Controlled Trial
Brief Title: Efficacy of Balloon-Expandable Stent Versus Self-Expandable Stent for the Atherosclerotic ILIAC Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seung Woon Rha, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENS-ILIAC
Record Dates: First submitted 2012-05-08; First posted 2013-04-18 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Artery Disease; Atherosclerosis
Keywords: Peripheral artery disease; atherosclerosis; stent
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balloon expandable stent (Experimental): study design is 1:1 randomization design. Patients will be randomized in a 1:1 manner according to different two (balloon expandable versus Self expandable)stents. Randomization procedure will be performed using a web-based program
  Interventions: Device: Balloon expandable stent
- Self expandable stent (Active Comparator): same to Balloon expandable stent
  Interventions: Device: Self expandable stent

INTERVENTIONS:
Device: Balloon expandable stent — provisional stenting should be performed; the case that optimal ballooning response in not obtained should be enrolled. Optimal balloon response is defined as a residual pressure gradient of > 15mmHg, residual stenosis of >30% and flow limiting dissection
  Other Names: SCUBA stent
  Arms: Balloon expandable stent
Device: Self expandable stent — provisional stenting should be performed; the case that optimal ballooning response in not obtained should be enrolled. Optimal balloon response is defined as a residual pressure gradient of > 15mmHg, residual stenosis of >30% and flow limiting dissection
  Other Names: COMPLETE SE
  Arms: Self expandable stent

SUMMARY:
The purpose of the investigators study is to examine and compare primary patency between balloon expandable cobalt chromium stent and self expandable nitinol stents (SCUBA versus COMPLETE-SE) in atherosclerotic iliac artery lesion.

DETAILED DESCRIPTION:
Obstructive atherosclerotic disease of the distal aorta and iliac arteries is preferentially treated with endovascular techniques, and an endovascular-first strategy can be recommended for all TransAtlantic Inter-Society Consensus (TASC) A-C lesions. Low morbidity and mortality as well as a >90% technical success rate justify the endovascular-first approach. Currently, In an attempt to improve outcomes, stent use has increased, and a number of studies favor iliac stenting over simple Percutaneous Transluminal Angioplasty (PTA). A meta-analysis comparing iliac stenting to Percutaneous Transluminal Angioplasty (PTA) found that stenting had higher rates of technical success and was associated with a 39% reduction in the risk of long-term loss of patency.

However, randomized control trial for comparison of primary patency between balloon expandable stent and self expandable stent has not been done, although there were some trials in that primary patency was compared among balloon expandable stents or among self expandable stents.

Currently, The choice of balloon versus self expandable stents is determined mainly by operator preference. The main advantages of balloon expandable stents are the higher radial stiffness and the more accurate placement, which is especially important in bifurcation lesions. In the external iliac artery, a primary stenting strategy using self-expandable stents compared with provisional stenting is preferred mainly due to a lower risk of dissection and elastic recoil.

Thus, the purpose of our study is to examine and compare primary patency between balloon expandable stent and self expandable stent(SCUBA versus COMPLETE SE stent)

ELIGIBILITY:
Inclusion Criteria:

1.Clinical criteria:

1. symptomatic peripheral-artery disease with

   * moderate to severe claudication (Rutherford 2-3),
   * chronic critical limb ischemia with pain while was at rest (Rutherford 4),
   * or chronic critical limb ischemia with ischemic ulcers (Rutherford 5-6)
2. Patients with signed informed consent

2. Anatomical criteria:

1. Target lesion length ≥ 4 cm by angiographic estimation,
2. Stenosis of more than 50% or occlusion of the ipsilateral iliac artery,
3. Patent (≤50% stenosis) ipsilateral femoropopliteal artery or concomitantly treatable ipsilateral femoropopliteal lesions (≤30% residual stenosis),
4. At least one patent (less than 50% stenosed) tibioperoneal runoff vessel.

Exclusion Criteria:

1. Disagree with written informed consent
2. Major bleeding history within prior 2 months
3. Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel or contrast agent
4. Acute limb ischemia
5. Untreated inflow disease of the distal aorta (more than 50 percent stenosis or occlusion)
6. Patients that major amputation ("above the ankle" amputation) has been done, is planned or required
7. Patients with life expectancy <1 year due to comorbidity
8. Age > 85 years

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-10-28 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Primary patency rate | 1year
  stenosis of at least 50 percent of the luminal diameter in the treated segment 12 months after intervention, as determined by quantitative angiography or CT angiography or peak systolic velocity ratio >2.5 by duplex sonography according to the stent type

SECONDARY OUTCOMES:
Clinical outcome | 1 year
  Limb salvage (free of above-the-ankle amputation)
Clinical outcome | 1 year
  Sustained clinical improvement rate at 12 month follow-up
Clinical outcome | 1 year
  Ankle-brachial index (ABI) at 12 months
Clinical outcome | 1 year
  The rate of major adverse cardiovascular events (MACE) at 12 months
Clinical outcome | 1year
  Repeated target lesion revascularization (TLR) rate
Angiographic outcome | 1 year
  Stent fracture rate
Angiographic outcome | 1 year
  Incidence of geographic miss
Clinical outcome | 1 year
  Repeated target extremity revascularization (TER) rate

CONTACTS AND LOCATIONS:
Overall Officials: Seung Woon Rha, MD. PhD, Principal Investigator — Cardiovascular center, Korea University Guro Hospital, 80, Guro-dong, Guro-gu, Seoul, 152-703, Korea
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi WG, Rha SW, Choi BG, Park S, Kim JB, Kang DO, Choi CU, Seo YS, Cho YH, Park SH, Lee SJ, Ko YG, Her AY, Kim SM, Kim KC, Cho JH, Kang WY, Kim JH, Kim MW, Kim DH, Bae JH, Ahn JH, Jo SC, Seo JB, Jung WY, Park SM; SENS-ILIAC Investigators. Balloon-expandable cobalt chromium stent versus self-expandable nitinol stent for the Atherosclerotic Iliac Arterial Disease (SENS-ILIAC Trial) Trial: a randomized controlled trial. Heart Vessels. 2024 Dec;39(12):1060-1067. doi: 10.1007/s00380-024-02431-4. Epub 2024 Jul 2. PMID 38953938
- [Derived] Choi WG, Rha SW, Choi CU, Kim EJ, Oh DJ, Cho YH, Park SH, Lee SJ, Hur AY, Ko YG, Park SM, Kim KC, Kim JH, Kim MW, Kim SM, Bae JH, Bong JM, Kang WY, Seo JB, Jung WY, Cho JH, Kim do H, Ahn JH, Kim SH, Jang JY; SENS-ILIAC Investigators. Study design and rationale of the 'Balloon-Expandable Cobalt Chromium SCUBA Stent versus Self-Expandable COMPLETE-SE Nitinol Stent for the Atherosclerotic ILIAC Arterial Disease (SENS-ILIAC Trial) Trial': study protocol for a randomized controlled trial. Trials. 2016 Jun 25;17(1):302. doi: 10.1186/s13063-016-1435-9. PMID 27344435